CLINICAL TRIAL: NCT05330832
Title: Covid-19 Associated Coagulopathy Predicted by Thrombodynamic Markers (CoViTro-I)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Other Study IDs: NCHPOI-2021-11
Record Dates: First submitted 2022-02-22; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-01

CONDITIONS: Coronavirus Disease 2019
Keywords: COVID-19; venous thromboembolism; pulmonary embolism; myocardial infarction; ischemic stroke; atherothrombosis
MeSH Terms: conditions — COVID-19; Venous Thromboembolism; Pulmonary Embolism; Myocardial Infarction; Ischemic Stroke; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood (Ailiton, UNIVAC plastic tubes, 4,5 mL with Sodium citrate 3,2%)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with confirmed SARS-Cov-2 infection: Hospitalized patients with modern or critical condition with confirmed COVID-19 infection. Patients received standard therapy for COVID-19 infection and anticoagulant prophylaxis if needed according to current temporary clinical recommendations.
  Interventions: Diagnostic Test: Thrombodynamics test

INTERVENTIONS:
Diagnostic Test: Thrombodynamics test — Thrombodynamics test is a global hemostasis test that allows to register the dynamics of fibrin clot formation in time and space. It requires whole blood samples from included patients.

SUMMARY:
The aim of the study is estimating the predictive and preventative capability of thrombodynamics for severe pneumonia coagulopathy complications in patients with COVID-19 infection. Thrombodynamics test is a method for blood coagulation and anticoagulation monitoring. It could be a useful tool for predicting thrombohemorrhagic complications in patients with COVID-19 infection and developing a novel scheme of anticoagulant therapy.

Inclusion criteria are the following: patient informed concern, confirmed COVID-19 diagnosis, state of modern or critical condition.

DETAILED DESCRIPTION:
The novel coronavirus viral infection (currently classified as COVID-19) causes a significant increase in death rate worldwide. Most of the patients with COVID-19 develop respiratory failure as well as coagulopathy.

The International Society of Thrombosis and Hemostasis (ISTH) has recently published guidelines for the treatment of coagulopathies in patients with COVID-19. It suggests using prophylactic doses of low molecular weight heparin (LMWH) in all patients with COVID-19. Numerous studies show a high percentage of thromboembolic complications in patients with COVID-19 as well as its potential association with pulmonary vessels microthrombosis and the development of acute respiratory distress syndrome. It is believed that COVID-19-associated coagulopathy could happen presumably due to the systemic inflammation. However, there are still no unified criteria for anticoagulant prophylaxis in such patients.

What is more, the severity of COVID-19 infection is also associated with high risk of life-threatening conditions such as sepsis and disseminated intravascular coagulation syndrome with massive uncontrolled bleeding.

According to the current clinical guidelines, coagulopathy in COVID-19 can be only registered with standard tests (prothrombin time (PT), platelet concentration and D-dimer). However, the lengthening of PT and the drop in platelet concentration are useful for the indication of the consumption stage of DIC. These changes mean that any patient remains already at risk of bleeding and the LMWH is no longer effective. The concentration of D-dimers shows the lysis of clots formed as a result of hypercoagulation, which also makes it a "delayed" marker of hypercoagulation. Thus, there are currently no reliable laboratory tools for hypercoagulation diagnostics in patients with COVID-19.

Thrombodynamics test is a global hemostasis test that allows to register the dynamics of fibrin clot formation in time and space. This test is highly sensitive to both hyper- and hypocoagulation and, at the same time, it allows to control anticoagulant therapy with heparins. The use of thrombodynamics test for the prediction of thrombohemorrhagic complications in this group of patients could be useful for individual correction of anticoagulant treatment and prevention of coagulopathy in COVID-19.

The aim of the study is estimating the predictive capability of thrombodynamics for SARS-CoV-2 associated coagulopathy in patients with severe pneumonia.

ELIGIBILITY:
Inclusion Criteria:

1. Patient (or the health care surrogate) Informed consent
2. Confirmed COVID-19 diagnosis

Exclusion Criteria:

1) Patient (or the health care surrogate) refusal to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of hospitalized patients with confirmed COVID-19 infection from April till December 2020 from 5 Moscow hospitals #40, 51, 23, 64 and the Troitsk hospital.
Sampling Method: Probability Sample
Enrollment: 2200 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2022-04-21 (Estimated)

PRIMARY OUTCOMES:
OS | From study enrollment until the date of death from any cause, assessed up to 4 months
  Outcome Measure - In-hospital mortality rate

SECONDARY OUTCOMES:
Myocardial infarction | 4 months from study enrollment
  Percentage of patients with in-hospital myocardial infarction
Ischemic stroke | 4 months from study enrollment
  Percentage of patients with in-hospital ischemic stroke
Arterial thrombosis | 4 months from study enrollment
  Percentage of patients with in-hospital arterial thrombosis
Venous thromboembolism, | 4 months from study enrollment
  Percentage of patients with in-hospital venous thromboembolism
DVT | 4 months from study enrollment
  Percentage of patients with in-hospital disseminated intravascular coagulation
Percentage of patients in moderate condition with in-hospital clinical deterioration | 4 months from study enrollment
  (respiratory rate > 30 per minute, SpO2 ≤ 93%, PaO2 /FiO2 ≤ 300 mm Hg, CT chest findings of the increase in the area of infiltrative changes for more than 50% in 24-48 hours, respiratory support necessity, unstable hemodynamics, multiple-organ-failure syndrome, qSOFA score > 2, arterial blood lactate > 2 mmol)
Percentage of patients in moderate critical with in-hospital clinical deterioration | 4 months from study enrollment
  (respiratory support necessity, unstable hemodynamics, multiple-organ-failure syndrome, qSOFA score > 2, arterial blood lactate > 2 mmol)

CONTACTS AND LOCATIONS:
Locations (1):
- Dmitry Rogachev National Medical Research Centre of Pediatric Hematology, Oncology and Immunology, Moscow, Russia